CLINICAL TRIAL: NCT02466321
Title: Anatomical Shoulder™ Inverse/Reverse Post-Market Surveillance Study
Brief Title: Anatomical Shoulder™ Inverse/Reverse Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer, GmbH (Industry)
Responsible Party: Sponsor
Organization: Zimmer Biomet (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-U02
Record Dates: First submitted 2015-06-03; First posted 2015-06-09 (Estimated); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-02

CONDITIONS: Cuff-tear Arthropathy
Keywords: Inverse Reverse Shoulder
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Inverse / Reverse Shoulder (Experimental): Patient treated with a inverse / reverse shoulder device.
  Interventions: Procedure: Inverse/Reverse Shoulder Arthroplasty

INTERVENTIONS:
Procedure: Inverse/Reverse Shoulder Arthroplasty — Implantation of the Anatomical Shoulder Inverse/Reverse System

SUMMARY:
The purpose of this study is to obtain outcomes data on the Anatomical Shoulder™ Inverse/Reverse System by analysis of standard scoring systems and radiographs.

Outcome data will be collected using the following standard scoring systems of which summary statistics will be provided:

• Constant and Murley Score to evaluate clinical parameters such as range of motion, power, level of pain and functional ability.

DETAILED DESCRIPTION:
This is a multi-centre, non-comparative, prospective post-market surveillance study involving orthopaedic surgeons skilled in shoulder replacement surgery. Each case enrolled will receive an Anatomical Shoulder™ Inverse/Reverse implant. All system components are CE-marked and commercially available. Patients will be selected according to the subject selection criteria.

All patients will undergo pre-operative, intra-operative and post-operative physical examination, radiographic evaluation according to the hospital's routine procedure and collection of quality of life metrics. Follow-up evaluations are to be conducted at either 6 weeks or 6 months (according to the hospital's standard care plan) and thereafter at 1, 2, 5 and 10 years post hospital discharge.

There are 5 study centres taking part in this project enrolling in total a maximum of 160 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age - 18 years minimum.
* Sex - male and female.
* General Health - the patient should be able to undergo surgery and participate in a follow-up program based upon physical examination and medical history.
* Informed Consent - patient or patient's legal representative has signed a Patient Informed Consent form.
* Indications - Diagnosis of disease or trauma in the affected joint, including cuff-tear arthropathy, failure of prior rotator cuff surgery and irreparable rotator cuff tears associated with loss of glenohumeral stability with the indication for total shoulder arthroplasty.
* The deltoid muscle has to be intact in all 3 parts (clavicular, acromial as well as spinal).

Exclusion Criteria:

* Patient is skeletally immature.
* Patient is pregnant.
* Patient is unwilling or unable to cooperate in a follow-up program.
* Patient shows one of the following medical conditions - Chronic fracture, Acute fracture, Axillary nerve lesion, Severe loss of humeral or glenoid bone, Paralysis of the deltoid muscle, Active Infection
* Patient requires one of the following medical interventions - Implant Revision, Glenoid bone grafting, Autografts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2007-05-16 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2024-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliott Goff, PhD, Study Chair — Zimmer Biomet, Jr. Clinical Project Lead
Locations (5):
- AZ Monica Antwerpen, Antwerp, Belgium
- Germany (2):
  - HELIOS ENDO-Klinik Hamburg, Hamburg
  - Vitos Orthopädische Klinik Kassel, Kassel
- Uniklinik Balgrist, Zurich, Switzerland
- The Pennine Acute Hospital NHS Trust, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Implants
Groups:
- Anatomical Shoulder Inverse/Reverse Prosthesis: Subjects implanted with the Anatomical Shoulder Inverse/reverse prosthesis
Period: Overall Study
Arm/Group | Anatomical Shoulder Inverse/Reverse Prosthesis
Started (Signed informed consent) | 154; 154 Implants (154 participants enrolled with signed informed consent. 153 patients operated (1 intention-to-treat-patient))
Received Study Device | 153; 153 Implants
Completed | 61; 61 Implants
Not Completed | 93; 93 Implants
Not completed — Death | 26
Not completed — Revision | 6
Not completed — Lost to Follow-up | 60
Not completed — Did not receive study device | 1

BASELINE CHARACTERISTICS:
Population: 154 participants were enrolled with signed informed consent whereas only 153 participants received the study device. 153 is the number that serves for the final analysis
Units Other Than Participants: implants
Arm/Group | Inverse / Reverse Shoulder
Number analyzed (Participants) | 153
Number analyzed (implants) | 153
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 153 is the number for the analysis
  years | 74.4 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 155 participants were enrolled, 153 serve as basis for the analysis
  Participants
    Female | 97
    Male | 56
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Number; unit: participants] — Population: 155 participants were enrolled, only 153 cases were operated with the study device and serve for the final results.
  participants
    Belgium | 19
    United Kingdom | 13
    Switzerland | 50
    Germany | 71
BMI [Mean (Standard Deviation); unit: kg/m2] — Population: 155 participants were enrolled but the analysis of results are based on 153 participants implanted with the study device
  kg/m2 | 27.2 (4.5)
Height [Mean (Standard Deviation); unit: cm] — 155 participants were enrolled but 153 participants that received the study device were included in the analysis Population: 153 is the number of participants receiving the study device , this number serves the final analysis
  cm | 165.0 (8.4)
Weight [Mean (Standard Deviation); unit: kg] — Population: 153 participants received the study device and serve as the final analysis
  kg | 74.1 (14.3)

OUTCOME MEASURES:

1. Primary Outcome: Functional Performance
Description: Constant & Murley Score. This evaluates clinical parameters such as range of motion, power, level of pain and functional ability. The score ranges from 0 - 100 with a higher score representing a better outcome.
Time Frame: 10 years
Population: For 42 participants constant & Murley score were available from baseline to 10 years follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Implants
Arm/Group | Inverse / Reverse Shoulder
Number analyzed (Participants) | 42
Number analyzed (Implants) | 42
score on a scale | 57.9 (15.8)

2. Secondary Outcome: Survival (Kaplan-Meier)
Description: The Kaplan-Meier estimator is a non-parametric statistic used to estimate the survival function from lifetime data. It is used to measure the fraction of patients living (in this case without a revision surgery) for a certain amount of time after treatment. A higher score is a better outcome.
Time Frame: 10 years
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | Inverse / Reverse Shoulder
Number analyzed (Participants) | 153
Number analyzed (Implants) | 153
Implants | 147

ADVERSE EVENTS:
Time Frame: AEs were collected from the time of surgery until study completion (up to 10 years)
Description: Seriousness of the Adverse Events were not assessed. Therefore, all Adverse Events are listed in the Serious Adverse Events table.
Arm/Group | Inverse / Reverse Shoulder
All-Cause Mortality (participants affected / at risk) | 26/153
Serious Adverse Events (participants affected / at risk) | 58/153
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inverse / Reverse Shoulder (N=153)
Death due to unrelated reasons (General disorders) | 26 (26)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Cardiac Arrhythmia (Cardiac disorders) | 2 (2)
Dislocation (Musculoskeletal and connective tissue disorders) | 2 (2)
Fracture of femoral neck (Musculoskeletal and connective tissue disorders) | 1 (1)
Fracture of proximal humerus (Musculoskeletal and connective tissue disorders) | 5 (5)
Glenoid implant failure (Musculoskeletal and connective tissue disorders) | 1 (1)
Glenoid implant loosening (Musculoskeletal and connective tissue disorders) | 3 (3)
hematoma (Blood and lymphatic system disorders) | 2 (2)
hemorrhage (Blood and lymphatic system disorders) | 1 (1)
humeral implant loosening (Musculoskeletal and connective tissue disorders) | 1 (1)
Nerve deficit (Nervous system disorders) | 1 (1)
nerve injury (Nervous system disorders) | 1 (1)
Other general complication (not shoulder) (General disorders) | 16 (16)
Other shoulder related complication (Musculoskeletal and connective tissue disorders) | 4 (4)
respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wound dehiscence (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-02-20): https://cdn.clinicaltrials.gov/large-docs/21/NCT02466321/Prot_SAP_000.pdf